CLINICAL TRIAL: NCT07191665
Title: Exploring Cortical Oxygenation Modulations in Response to Dietary Components During Cognitive Activity in Healthy Adults: a fNIRS Study
Brief Title: Explore the Use of Cortical Oxygenation Measures in Nutrition Research
Acronym: Saga
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Other Study IDs: 2305NR
Record Dates: First submitted 2023-12-07; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Functional Near Infrared Spectroscopy; Cortical tissue oxygenation; Cognition; Mental fatigue; Workload; Caffeine; L-Arginine
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy males and females aged between 25 and 35 years old.
  Interventions: Other: Acute nutrition intervention

INTERVENTIONS:
Other: Acute nutrition intervention — The products (investigational and placebo) consists of three capsules that should be taken with water at two separate visits, with a wash-out period in between. The placebo product will comprise of microcrystalline cellulose (bulk). The investigational products will contain either caffeine and microcrystalline cellulose or caffeine, L-Arginine, and microcrystalline cellulose.

SUMMARY:
The current project aims to explore the use of cortical oxygenation measures obtained with functional Near Infrared Spectroscopy (fNIRS) in acute nutrition interventions with outcomes on cognition.

DETAILED DESCRIPTION:
The project aims to test a previously developed fNIRS-based protocol for evaluating the acute effects of dietary components on cognitive function in a population of healthy young adults. The testing will involve detecting patterns in fNIRS-based cortical tissue oxygenation level and cognitive performance that are expected due to the bioactive mechanisms of the studied components.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 25-35 years old
* BMI between 18.5 kg/m2 and 29.9 kg/m2
* Conditions for study procedure compliance:

  * Willing and able to sign an informed consent form
  * Fluent in English (self-reported C1 or C2 English level)
  * Have reliable cortical oxygenation signal for subsequent analysis (based on the real-time computation of a parameter reflecting the quality of the signal, which may be influenced by variations in hair thickness)
  * Dominant right-handed
  * Have normal or corrected-to-normal vision
  * Willing and able to comply with the protocol requirements

Exclusion Criteria:

* Conditions that may affect cortical oxygenation:

  * Have a past or current neural, cerebrovascular, cardiovascular, or respiratory disease (based on anamnesis)
  * Have a past or current kidney disease or condition (based on anamnesis)
  * Measured hypo- or hyper-tension (verified by evaluating Blood Pressure, BP, measure against medical norms at screening)
  * Self-reported, suspected or diagnosed migraine (based on anamnesis)
  * Have a mild or clinical form of insomnia (verified by thresholding rated insomnia severity index, ISI, at or above 8) or being a night shift worker (based on anamnesis)
  * Regular smoker, regularly is being defined as more than 2 cigarettes per week
  * Participating in vigorous physical activity defined as requiring more than 6 metabolic equivalents (e.g., hiking, jogging at 10 km/h or more, carrying of heavy loads, bicycling fast at 23 km/h or more, basketball, soccer, and tennis single), greater than 4 times 45 minutes per week
* Conditions that may affect cognition or mental fatigue:

  * Have a current psychiatric disorder or have a self-reported, suspected or diagnosed anxiety or depression (based on anamnesis)
  * Taking illicit drugs for e.g., cannabis, heroin, and cocaine
  * Have an average alcohol consumption defined as greater than 2 standard drinks per day over a week for males, and greater than 1 standard drink per day over a week for females. One standard drink contains 10-12 g of ethanol. Examples of standard drinks are one beer can (300 ml), one glass of wine (100 ml) or one glass of schnaps (30 ml).
  * Pregnant (verified by a pregnancy test in urine dipstick format provided by the study's site) or seeking to become pregnant or breast feeding (based on anamnesis)
* Conditions that may interact with the IP mechanism:

  * Have food allergies and intolerances (based on anamnesis)
  * Have a high usual consumption of caffeine-based beverages and foods (verified by thresholding the daily consumption of caffeine as determined by the Caffeine Consumption Questionnaire, CCQ, at or above 600mg)
  * Body mass below 60kg (associated with a dosing of more than 3mg caffeine per 1kg of body mass)
  * Currently taking Sildenafil (based on anamnesis)
  * Self-reported, suspected or diagnosed with acute inflammatory diseases e.g., herpes simplex virus, allergies, or asthma (based on anamnesis)
* Have a hierarchal or family relationship with any of the research team members.
* Currently participating in an interventional study.

Ages: 25 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: The study population will comprise of 36 healthy adults from 25 to 35 years old. To analyze gender-related differences, the population will be equally distributed according to gender.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Caffeine-induced pattern of correlation between cortical tissue oxygenation and cognitive performance (relative to placebo). | Change in correlation from baseline to 45' post-product intake ; This measurement is performed for each product. Each product is given a single time. 5-9 days between each of the products assigned.
  Detect a pattern of correlation between caffeine-induced changes in cortical tissue oxygenation and cognitive performance. Cognitive performance will be assessed using accuracy and reaction time data collected from cognitive tests, such as memory tests.
Caffeine-induced pattern of correlation between cortical tissue oxygenation and cognitive performance (relative to placebo) | Change in correlation from baseline to 45' post-product intake ; This measurement is performed for each product. Each product is given a single time. 5-9 days between each of the products assigned.
  Detect a pattern of correlation between caffeine-induced changes in cortical tissue oxygenation and cognitive performance. Cortical tissue oxygenation level will be measured by analyzing changes in oxygenated or deoxygenated hemoglobin concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Pamela, Medical, Principal Investigator — Société des Produits Nestlé
Locations (1):
- Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Access to the data will only be given to the academic laboratory hosting the the aforementioned doctoral study. This concerns the Medical Image Processing laboratory, Ecole Polytechnique Fédérale de Lausanne.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will only be available from the preliminary to the last analysis performed (i.e. end of the study).
Access Criteria: A thesis agreement to cover the data protection has been agreed with the laboratory of the doctoral thesis director. The access to the data will be performed via secure directories of Société des Produits Nestlé.